CLINICAL TRIAL: NCT01979224
Title: Efficacy of Educational Intervention for Parents of Children With Asthma in 4-11 Years and Their Impact on the Control Children as Measured by ACT. Randomized Controlled Clinical
Brief Title: Efficacy of Educational Intervention for Parents of Children With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Collaborators: Hospital General de Soledad de Graciano Sánchez, SLP, MX (Unknown)
Responsible Party: Principal Investigator, Blanca Nohemí Zamora Mendoza, Efficacy of educational intervention for parents of children with asthma in 4-11 years and their impact on the control as measured by childern Asthma Control Test (ACT). Randomized Controlled Clinical, Universidad Autonoma de San Luis Potosí
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-001; UASLP-001 (Registry Identifier: UASLP-001)
Record Dates: First submitted 2013-05-30; First posted 2013-11-08 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-10

CONDITIONS: Asthma
Keywords: educational intervention, Asthma control, asthma knowledge
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment and routine counseling (No Intervention): Parents attend regular consultation and receive regular medical guidance
  Interventions: Other: Educational intervention for parents

INTERVENTIONS:
Other: Educational intervention for parents — educational sessions once a week two hours for a month and later educational reinforcement and monitoring asthma control monthly for nine months
  Other Names: Educational intervention for parents of children with asthma

SUMMARY:
Introduction. Asthma is a chronic inflammatory disorder of the airways, identified by airflow obstruction. Unfortunately only 2.4% of American asthmatics meet internationally recommended criteria for control. The lack of knowledge in parents of asthmatic children has been a direct result of minimum or no control at all, so the educational programs need to be assessed in terms of improvement of the control. Target. To determine whether an educational intervention aimed at parents of asthmatic children 4 to 11 years improved clinical control measured by Test Childhood Asthma Control. Material and Methods. Randomized controlled clinical trial in 42 patients randomly divided into two groups that were evaluated in the same time knowledge and control of asthma, a measurement was performed at baseline and monthly for nine months. The experimental group attended an educational intervention for individual reinforcements through this period, the control group was only monitored

DETAILED DESCRIPTION:
* Recruitment of patients that attended hospital's emergency gate due to asthma issues, and phone calls to regular physicians patients.
* Once recruited all parents of patients were asked to participate in the study where their children will be evaluated on an asthma control and asked informed consent
* The clinical history, spirometry and / or basal peak flow Diagnostic concordance
* With the collected data was performed a database clinical history, ACT score, FEV1 and PEF, results of each patient and personal data for future location, the base was used for the concordance of diagnosis.
* Once the sample that met the selection criteria were formed experimental and control groups at random using "R Project Statistical Computing" 2.12.2 version performed by the statistical
* The experimental group was invited to participate in educational sessions two hours at week in just one month and monthly individual reinforcements through the evaluation period.
* Educational sessions were based on the Global Initiative for Asthma (GINA), Guía Española para el Manejo del Asma (GEMA) And Concenso Mexicano de Asma.
* Those measurements were performed by an external partner or educators or the attending physician performed to avoid biased results.

The monthly ACT and peak flow of the attending physician were blinded

variables:

* educational intervention, with and without intervention
* asthma control: measured by infant ACT
* time: 0 to 9 months
* sex: female or male
* Age: 4 to 11 years

ELIGIBILITY:
Eligibility Criteria

* Children 4-11 years with diagnosed asthma with parents attending the outpatient pediatric pneumology and pediatric emergency because of acute asthma in General Hospital de Soledad.
* Patients with a baseline score less than 27 points in childhood ACT
* Patients with Government Health Insurance. (to ensure access to medication and medical care)
* Parents who can read and write
* Parents willing and able to participate
* Parents who do not belong or have been part of an educational program on asthma by asthma clinic.

Exclusion Criteria

- Parents with children having other comorbidities that prevent or hinder proper control of asthma, such as Cerebral Palsy, (PCI) psychomotor retardation, psychiatric Sd. Down, congenital malformations, which alter the chest wall, obesity, nasal polyp.

Elimination criteria

* Parents who fail to attend 50% of the sessions given (since it does not allow parents to acquire sufficient knowledge to significantly improve the control of asthma as GEMA educational guidance)
* Patients and parents who decide not to continue in the project.
* Patients who develop pulmonary comorbidities over a month of evolution and lung tissue affecting significantly, as syncytial respiratory virus, pneumonia, tuberculosis, and asthma control difficulties.
* Patients who leave or do not take the prescribed treatment by physician for a month.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
asthma control | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Blanca ZM master, Principal Investigator — Universidad Autónoma de San Luis Potosí México